CLINICAL TRIAL: NCT02126293
Title: Correction of Zinc Deficiency in Children With Chronic Kidney Disease and Kidney Transplant
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: London Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZICKD13-827
Record Dates: First submitted 2014-01-30; First posted 2014-04-30 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Renal Insufficiency, Chronic; Zinc Deficiency; Trace Element Excess; Trace Element Deficiency
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Urinalysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Zinc deficient patients (Experimental): If the patient is found to be zinc deficient (serum zinc < 11.5 μmol/L), the family will be contacted by the RA to commence zinc supplement: zinc citrate (Zinc Lozenges, manufactured by Douglas Laboratories Inc, London, ON, Health Canada NPN 80032476) for 3 months. As per the NPN licence the dose is 10 mg (1 lozenge) orally once a day for children age 4-8 years, and 10 mg twice a day for children age 9-18 years. This should give enough time to restore serum zinc to normal in most patients.
  Interventions: Drug: Zinc Supplement
- Zinc sufficient patients (Active Comparator): Zinc sufficient patients will repeat blood and urine tests in 3 month time to compare the changes with intervention arm.
  Interventions: Procedure: Repeat blood and urine tests

INTERVENTIONS:
Drug: Zinc Supplement
  Other Names: Zinc Lozenges,Douglas Laboratories,HC NPN 80032476
  Arms: Zinc deficient patients
Procedure: Repeat blood and urine tests
  Arms: Zinc sufficient patients

SUMMARY:
Children with chronic kidney disease, even after transplantation, may be at risk for bone problems due to an imbalance of calcium and phosphorus in the blood, especially as their kidneys progressively fail to function. While some drug and diet treatments are available to prevent such bone disease, many children refuse to take them due to bad taste and tummy cramps. If calcium and phosphorus status remain abnormal for a long time, hard crystals can form in the blood vessels, eventually clogging them and resulting in heart problems. Investigators are studying possible new methods to help the kidneys maintain a normal balance of nutrients in the blood which is important for growing healthy bones and the prevention of side effects in blood vessels that can lead to heart disease. One method is to improve the team work of a hormone FGF-23 and a protein called Klotho that together stimulate the kidneys to increase phosphate removal. Investigators propose that this problem may be due to low blood zinc levels which often occur in children with kidney disease. Thus, in this study, investigators propose to first measure zinc in blood from children with chronic kidney disease (CKD) or who have had kidney transplants to assess zinc and phosphate status, the hormone FGF-23 and its assistant Klotho. If zinc status is low, the children will receive zinc supplementation for 3 months. After treatment with zinc, the same blood measurements will be repeated to determine if the zinc supplements have helped the hormones to remove phosphate from the body. If this pilot project is successful, investigators will then consider a larger scale project involving adult patients as well as pediatric patients from other pediatric centers. This project will also guide investigators as to whether they need to introduce zinc measurements as part of routine testing of CKD and transplant patients. In addition to measuring zinc levels in study participants, trace elements (TE) will also be measured. These include heavy metals such as cadmium, chromium, nickel, vanadium, copper, lead, manganese and selenium. Very little is known about levels and metabolism of TE in CKD especially before dialysis. In adults, cadmium, chromium, nickel, and vanadium probably accumulate in hemodialysis patients, while copper and lead may accumulate. Manganese, selenium are probably deficient. The study will allow investigators to obtain the information about TE in this group of pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Children between 4 and 18 years of age; diagnosis of CKD; renal transplant recipient with declining renal function (eGFR<90 ml/min/1.73 m2).

Exclusion Criteria:

* Children with CKD or kidney transplant younger than 4 years. Kidney transplant recipients with eGFR>90 ml/min/1.73 m2.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Establish proportion of zinc deficient children with chronic kidney disease and kidney transplant, who achieved correction of zinc deficiency after 3 months of zinc therapy | 3 months of therapy

SECONDARY OUTCOMES:
Change in parameters of bone metabolism following zinc treatment in zinc deficient patients | Baseline and 3 months
  Correlations between various parameters of bone metabolism, kidney function, zinc, FGF-23 and Klotho assessed by a multiple regression model. Change from baseline in FGF-23, Klotho, TE levels and phosphate excretion after zinc therapy analyzed by a paired t-test.
TE levels in zinc deficient children with chronic kidney disease and kidney transplant | Baseline and 12 weeks
  Establish TE levels in zinc deficient children with chronic kidney disease and kidney transplant. Establish changes in TE levels following correction of zinc deficiency.
TE levels in zinc sufficient children with chronic kidney disease and kidney transplant | Baselne and 12 weeks
  Establish TE levels in zinc sufficient children with chronic kidney disease and kidney transplant. Establish TE levels 12 weeks later as a quality control measure.

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Belostotsky, MD, PhD (eq), Principal Investigator — Hamilton Health Sciences Corporation
Locations (2):
- Canada (2):
  - McMaster Children's Hospital, Hamilton, Ontario
  - Children's Hospital, London Health Science Centre University of Western Ontario, London, Ontario

REFERENCES:
- [Derived] Filler G, Taheri S, McIntyre C, Smith C, Subramanian L, Fusch G, Fusch C. Chronic kidney disease stage affects small, dense low-density lipoprotein but not glycated low-density lipoprotein in younger chronic kidney disease patients: a cross-sectional study. Clin Kidney J. 2018 Jun;11(3):383-388. doi: 10.1093/ckj/sfx115. Epub 2017 Oct 12. PMID 29992019
- [Derived] Filler G, Kobrzynski M, Sidhu HK, Belostotsky V, Huang SS, McIntyre C, Yang L. A cross-sectional study measuring vanadium and chromium levels in paediatric patients with CKD. BMJ Open. 2017 Jun 6;7(5):e014821. doi: 10.1136/bmjopen-2016-014821. PMID 28592575